CLINICAL TRIAL: NCT05724901
Title: A Wearable Remote Data Capture Solution for Home-Based Gait Assessment in Multiple Sclerosis
Brief Title: At-Home Gait Assessment
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 22-00375
Record Dates: First submitted 2023-02-03; First posted 2023-02-13 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis
Keywords: Gait Analysis; telehealth; sensor-based gait analysis; home-based
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with MS: Participants will complete an in-clinic visit (self-reported outcome of MS disability, a standard walking clinical evaluation, and a sensor-based gait evaluation) and 3 remote supervised self-administered gait assessments using the MS-GRCA system.

SUMMARY:
The goal of this study is to validate an MS Gait Remote Capture and Analysis (MS-GRCA) system based on wearable shoe-based motion sensors for home-based and repeatable gait assessments.

DETAILED DESCRIPTION:
This is a single-site observational longitudinal study to validate an MS Gait Remote Capture and Analysis system for home-based and repeatable gait assessments. The investigators will recruit 30 participants who will have an in-person baseline visit (informed consent, standard gait assessment, sensor-based gait assessment, self-reported questionnaires), followed by three remote visits (sensor-based gait assessment, SUS questionnaire [last remote visit only]).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70 years old (inclusive)
* Confirmed diagnosis of MS (any MS subtypes, Relapsing Remitting [RR], Primary Progressive [PP], or Secondary Progressive [SP])
* PDSS score from 0 to 5
* Stable and continuous access to internet at home
* Adequate home facilities (enough space, quiet and distraction free area)
* Ability to provide informed consent.

Exclusion Criteria:

* Below average estimated premorbid cognitive functioning (based on WRAT-4 reading recognition standard z-score < 85).
* Presence of severe cognitive impairment (based on SDMT age normative z-score < -3.0).
* Presence of primary neurological disorders other than MS or primary psychiatric disorder that would influence ability to complete assessments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (ages 18-70) diagnosed with MS, any subtypes (Relapsing Remitting, Primary Progressive, or Secondary Progressive MS).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Mean Gait Velocity | Up to Week 4
  Measured using sensor-based gait assessment

SECONDARY OUTCOMES:
Mean Stride Length | Up to Week 4
  Measured using sensor-based gait assessment at baseline and remote visits 1, 2 and 3.
Mean Double Support Duration | Up to Week 4
  Double support duration represents the time that both feet are on the ground while walking. Measured using sensor-based gait assessment at baseline and remote visits 1, 2 and 3.
Mean Stance Duration | Up to Week 4
  Stance duration represents the duration of the time between heel strike and toe off of the same foot. Measured using sensor-based gait assessment at baseline and remote visits 1, 2 and 3.
Mean Cadence | Up to Week 4
  Cadence defined as number of steps per minute. Measured using sensor-based gait assessment at baseline and remote visits 1, 2 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT05724901/ICF_000.pdf